CLINICAL TRIAL: NCT02557048
Title: Malignant Head and Neck Tumors in Children: A Retrospective Study
Brief Title: Head and Neck Cancer in Children: A Retrospective Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohammed Morsy, MD, Lecturer, Pediatric Oncology Department, Assiut University
Other Study IDs: Ped Head Neck Malig
Record Dates: First submitted 2015-09-21; First posted 2015-09-22 (Estimated); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Head and Neck Neoplasms; Cancer of Head and Neck; Cancer of the Head and Neck; Head and Neck Cancer; Neoplasms, Head and Neck
Keywords: Childhood Cancer; Head and Neck Tumors; Pediatric Oncology
MeSH Terms: conditions — Head and Neck Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the study is to identify demographic characteristics, various histopathologies, and site preferences for each disease entity of malignant head and neck tumors in pediatric oncology patients & treatment outcomes in these patients, according to experience at South Egypt Cancer Institute which is the largest referral site in Upper Egypt.

DETAILED DESCRIPTION:
Background:

Although head and neck masses represent a common entity in children, malignancy is uncommon. Only very limited data are available in the literature on the incidence of childhood cancer of the head and neck worldwide.

Data from the United States National Cancer Institute database suggest that the head and neck are involved in 12 % of all childhood malignancies. The most common pediatric head and neck malignancies include Non Hodgkin lymphomas, Hodgkin lymphomas, rhabdomyosarcomas, thyroid malignancies, nasopharyngeal carcinomas (NPCs), salivary gland malignancies, and neuroblastomas.

Patients & Methods:

A hospital-based study, involving Pediatric cancer patients, those diagnosed with malignant tumors of the head & neck, in the period from 2001 January till 2015 December, and received treatment at the pediatric oncology department, their medical records will be retrospectively reviewed for data collection.

Clinico-laboratory data for each hisopathologic disease entity of various head & neck malignancies will be gathered. The demographic distribution for each disease entity in accordance with gender & age, and site preferences in these disease entities will be recorded. Treatment received & treatment outcomes will be verified and absolute frequencies & relative incidence of these disease entities will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose age less than 19 years.
* Patients diagnosed with a primary malignant tumor of the head & neck.

Exclusion Criteria:

* Patients whose age more than 18 years.
* Patients diagnosed with a malignant disease primarily arising from the bone marrow.
* Patients diagnosed with tumors of the central nervous system.
* Patients diagnosed with retinoblastoma.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: A hospital-based study, involving Pediatric cancer patients, those diagnosed with malignant tumors of the head & neck, in the period from 2001 January till 2015 December, and received treatment at the pediatric oncology department, their medical reports will be retrospectively reviewed for data collection.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2019-01-10 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | Participants will be retrospectively followed forward in time from the date of initiation of treatment till the primary completion date of the study, an expected average of 5 years
  Time from the date of initiation of treatment until death from any cause
Event Free Survival (EFS) | Participants will be retrospectively followed forward in time from the date of initiation of treatment till the primary completion date of the study, an expected average of 5 years
  Time from the date of initiation of treatment until disease progression, or death for any reason.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

REFERENCES:
- [Background] Chadha NK, Forte V. Pediatric head and neck malignancies. Curr Opin Otolaryngol Head Neck Surg. 2009 Dec;17(6):471-6. doi: 10.1097/MOO.0b013e3283323893. PMID 19745735
- [Background] Gosepath J, Spix C, Talebloo B, Blettner M, Mann WJ. Incidence of childhood cancer of the head and neck in Germany. Ann Oncol. 2007 Oct;18(10):1716-21. doi: 10.1093/annonc/mdm278. Epub 2007 Jul 28. PMID 17660492